CLINICAL TRIAL: NCT04848298
Title: Use of mHealth to Increase Physical Activity for Patients Recently Hospitalized With Acute Heart Failure: a Randomized Clinical Trial
Brief Title: Use of mHealth to Increase Physical Activity for Patients Recently Hospitalized With Acute Heart Failure
Acronym: mRehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IIBSP-MRE-2020-86
Record Dates: First submitted 2021-04-08; First posted 2021-04-19 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Health Arm (Experimental)
  Interventions: Behavioral: mHealth Intervention
- Control Arm (No Intervention): The Control Arm will receive standard of care including tailored prescription of physical activity

INTERVENTIONS:
Behavioral: mHealth Intervention — The Mobile Health Arm will receive standard of care including tailored prescription of physical activity as well as the mobile health intervention, which will have the following features:
  * Goal setting for frequency and duration of exercise sessions
  * Graphic feedback and reinforcement with educational and motivational messages tailored to user's exercise adherence.
  * Problem-solving support
  * Library with educational tips and information regarding physical exercise.
  Arms: Mobile Health Arm

SUMMARY:
The aim of this trial is to determine if a mobile application that promotes physical exercise in the follow-up of patients recently hospitalized with acute heart failure can improve exercise capacity after 6 months and physical activity levels compared to the standard follow-up.

A randomized clinical trial will be conducted with 100 consecutive patients aged +18 years, hospitalized for acute decompensated heart failure in a tertiary referral hospital who own a mobile phone compatible with MyPlan and access to Wi-Fi or mobile data. At discharge, patients will be randomly assigned in two groups; the intervention group will be followed with a smartphone application to promote physical activity, whereas the control group will take responsibility in their adherence to exercise recommendations. Main study variables will be functional capacity after 6 months, which will be evaluated using the six minute walking test, and physical activity levels, using the International Physical Activity Questionnaire (IPAQ). The study will be analyzed using the intention-to-treat principle. The project has been authorized by the local committee for ethics in clinical research.

ELIGIBILITY:
Inclusion Criteria:

* Aged +18 years
* Hospitalized for acute decompensated heart failure in a tertiary referral hospital
* Owning a mobile phone compatible with MyPlan and access to Wi-Fi or mobile data (either the patient or the caregiver)

Exclusion Criteria:

* NYHA IV patients
* Currently listed for heart transplant
* Left ventricular assist device recipient
* Ventricular arrhythmia within prior 6 months
* Uncontrolled arterial hypertension or resting heart rate >100 bpm
* Acute myocarditis or pericarditis
* Severe aortic stenosis
* Hypertrophic obstructive cardiomyopathy
* Advanced AV block
* Muscle-skeletal or neurologic disease preventing to perform study procedures
* ACS within prior month
* Severe lung disease
* Moderate or severe cognitive impairment
* Unable/unwilling to consent
* Projected life expectancy <6 months
* Clinical judgment concerning other safety issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Change in 6-minute walking distance (6MWD) | 6 months

SECONDARY OUTCOMES:
Participant reported physical activity levels, using the International Physical Activity Questionnaire (IPAQ) | 6 months
  Results will be reported in categories (low activity levels, moderate activity levels or high activity levels) and as a continuous variable (MET minutes a week)

OTHER OUTCOMES:
Muscle strength - measured using the Medical Research Council (MRC) Sum Score | 6 months
  The total MRC sum score ranges from 0 (total paralysis) to 60 (normal strength).
Upper limb strenght - measured by hand-held dynamometry | 6 months
  This instrument is scored using force production in kilograms (0-90)
Rectus femoris muscle diameter | 6 months
Physical function measured by the Short Physical Performance Battery score | 6 months
  Each task is scored from 0 to 4, with 4 being the best, and a total battery score of 12 points
Participant reported quality of life - measured using the Minnesota living with heart failure questionnaire (MLHFQ) | 6 months
  Each item is scored in a 6-point Likert Scale (0 to 5), thus the total score could range from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life
NT-proBNP levels | 6 months
Readmission rate for Heart Failure | 6 months
Participant reported time dedicated to exercise recommendations | 6 months
Number of steps -measured using the built-in smartphone pedometer | 6 months
User satisfaction with the mHealth application (only experimental arm), measured by a customer satisfaction survey specifically designed for the trial | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Mirabet, Ph. D., Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain